CLINICAL TRIAL: NCT01741363
Title: Screening for Stomach Diseases and Colorectal Neoplasms With the Fecal Testing: a Population-based Randomized Study
Brief Title: Screening for Stomach Diseases and Colorectal Neoplasms With the Fecal Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201205030RIB
Record Dates: First submitted 2012-10-05; First posted 2012-12-04 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer; Stomach Disease
Keywords: iFOBT; one-day sample; two-day sample; Helicobacter pylori stool antigen
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- one-day sampling with one-year interval (Experimental): FIT one-day sampling with one-year interval
  Interventions: Other: FIT(Eiken OC-Sensor) One-year interval; Other: FIT(Eiken OC-Sensor) One-day sampling
- one-day sampling with two-year interval (Active Comparator): FIT one-day sampling with two-year interval
  Interventions: Other: FIT(Eiken OC-Sensor) One-day sampling; Other: FIT(Eiken OC-Sensor) Two-year interval
- two-day sampling with one-year interval (Experimental): FIT two-day sampling with one-year interval
  Interventions: Other: FIT(Eiken OC-Sensor) Two-day sampling; Other: FIT(Eiken OC-Sensor) One-year interval
- two-day sampling with two-year interval (Experimental): FIT two-day sampling with two-year interval
  Interventions: Other: FIT(Eiken OC-Sensor) Two-day sampling; Other: FIT(Eiken OC-Sensor) Two-year interval
- Hp stool antigen (HpSA)+FIT (Experimental): HpSA for detection of upper gastrointestinal tract diseases and upper endoscopy for H. pylori carriers; HPSA combined with FIT
  Interventions: Other: FIT(Eiken OC-Sensor) One-day sampling; Other: FIT(Eiken OC-Sensor) Two-year interval; Other: HpSA (Firstep Helicobacter pylori Antigen Rapid Test)
- FIT only (Active Comparator): HpSA + FIT compared with FIT alone
  Interventions: Other: FIT(Eiken OC-Sensor) One-day sampling; Other: FIT(Eiken OC-Sensor) Two-year interval; Other: FIT only

INTERVENTIONS:
Other: FIT(Eiken OC-Sensor) Two-day sampling — Collect two stool samples in two separate days
  Arms: two-day sampling with one-year interval; two-day sampling with two-year interval
Other: FIT(Eiken OC-Sensor) One-year interval — Screening with one-year interval
  Arms: one-day sampling with one-year interval; two-day sampling with one-year interval
Other: FIT(Eiken OC-Sensor) One-day sampling — One-day sampling
  Arms: FIT only; Hp stool antigen (HpSA)+FIT; one-day sampling with one-year interval; one-day sampling with two-year interval
Other: FIT(Eiken OC-Sensor) Two-year interval — Screening with two-year interval
  Arms: FIT only; Hp stool antigen (HpSA)+FIT; one-day sampling with two-year interval; two-day sampling with two-year interval
Other: HpSA (Firstep Helicobacter pylori Antigen Rapid Test) — HpSA for detection of upper gastrointestinal diseases; screen and treat for H. pylori infection. Upper endoscopy for H. pylori carriers. HPSA+FIT compared with FIT alone.
  Arms: Hp stool antigen (HpSA)+FIT
Other: FIT only — HPSA+FIT compared with FIT alone.
  Arms: FIT only

SUMMARY:
1. The abundant results from this trial will be helpful for assessing the feasibility of increasing stool sampling and shortening screening interval in population setting for lower and upper gastrointestinal tract lesions, their long-term effects, and the respective cost-effectiveness.
2. The study will evaluate the value of population-based screen and treatment for H. pylori infection when the HPSA is combined with the FIT.

DETAILED DESCRIPTION:
Growing body of evidences have shown that fecal immunochemical test (FIT) outperform guaiac fecal occult blood test (gFOBT) in terms of sensitivity, neoplasm detection rate and public participation. Though direct outcome evidence is still lacking for FIT, it is anticipated to have higher colorectal cancer (CRC) mortality and incidence reduction compared with gFOBT. In Taiwan, nation-wide CRC screening program has been launched since the year of 2004 ,which provides biennial FIT screening for adults aged 50 to 69 years. Currently available data from the Bureau of Health Promotion has shown a significant stage-shift effect, an early indicator of screening effectiveness, by this screening program.

Nevertheless, the aforementioned advantages of FIT, missed neoplasms and interval cancer still exists under the current one-day stool sampling method with biennial screening interval, which might affect the effectiveness of overall screening program. Increase the number of stool samples or shortening of screening interval may be helpful for early detection of clinically significant neoplasms but it remains unclear whether such an approach may lower the screenee compliance or public participation. Moreover, its impact on the demand of confirmatory colonoscopy and cost-effectiveness of the whole screening program is still largely unknown and need to be further investigated.

In this study, we firstly aim to randomly allocate screening attendee to one of the following four arms: one-day sampling with annual screening, one-day sampling with biennial screening, two-day sampling with annual screening, and two-day sampling with biennial screening. Participation rate, positive rates of FIT, detection rate for neoplasms, positive predictive value, and long-term outcome including cancer incidence and mortality will be calculated and compared among four groups.

Secondly, in the Taiwanese population, which is a typical presentation of Asian populations, although the incidence of colorectal cancer is rapidly increasing, Helicobacter pylori-related upper gastrointestinal pathologies remain highly prevalent, which may imply that mass screening solely based on FIT could be insufficient as significant upper GI pathologies can be missed. Since the FIT does not predict upper GI pathologies, the adjunct of an「Helicobacter pylori stool-antigen test (HpSA) 」 may be a potential candidate to realize a pan-detecting assay based on stool samples in a population in which both lower and upper GI lesions are equally prevalent. Therefore, in the present study, we will also evaluate the value of simultaneous FIT and HpSA test in the community-based mass screening. We invited subjects in a randomized study to receive the FIT or the FIT plus HPSA. Those who are tested positive for HPSA will receive upper endoscopic examination and anti-H. pylori treatment. For the short-term indicators, we will evaluate the participation rate and diagnostic yield when the HPSA is added. For the long-term indicators, we will compare the incidence and mortality of gastric cancer as well as complicated peptic ulcers.

To summary, this study includes two randomized trials:

1. To make a comparison between one-day sampling with annual screening, one-day sampling with biennial screening, two-day sampling with annual screening, and two-day sampling with biennial screening using FIT;
2. To make a comparison between FIT plus HpSA and FIT alone for screening.

Finally, the cost-effectiveness analysis will be also conducted using previously established Markov model of CRC natural history and stomach diseases (such as dyspepsia, peptic ulcer disease, and gastric cancer) using the results ascertained from this trial. The primary outcomes were gastric cancer incidence and mortality rates as well as colorectal cancer incidence and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 69 years average-risk subjects for FIT
* 50 to 69 years subjects for HpSA

Exclusion Criteria (for the FIT-based RCT):

* Subjects who are unwilling to participate
* Subjects ineligible for colonoscopy (for the one-day vs two day FIT screening)

Exclusion Criteria (for the FIT+HPSA vs. FIT-only RCT)

* Subjects with a history of total gastrectomy
* Pregnancy
* Subjects with severe illnesses
* Subjects with prior participation in the pilot program

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99314 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Mo Chiu, M.D., Ph.D., Principal Investigator — Department of Internal Medicine & Health Management Center; Yi-Chia Lee, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YC, Chiang TH, Chiu HM, Su WW, Chou KC, Chen SL, Yen AM, Fann JC, Chiu SY, Chuang SL, Chen YR, Chen SD, Hu TH, Fang YJ, Wu MS, Chen TH, Yeh YP; Collaborators of Taiwan Community-based Integrated Screening Group. Screening for Helicobacter pylori to Prevent Gastric Cancer: A Pragmatic Randomized Clinical Trial. JAMA. 2024 Nov 19;332(19):1642-1651. doi: 10.1001/jama.2024.14887. PMID 39348147
- [Derived] Lee YC, Chiang TH, Chiu HM, Wu MS, Yeh YP, Hsiu-Hsi Chen T; Collaborators of the Taiwan Community-Based Integrated Screening Group. Community-Based Gastric Cancer Screening Coupled With a National Colorectal Cancer Screening Program: Baseline Results. Gastroenterology. 2021 May;160(6):2159-2161.e4. doi: 10.1053/j.gastro.2021.01.008. Epub 2021 Jan 11. No abstract available. PMID 33444571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2014/04/01 First patient first visit
Pre-assignment Details: 2018/09/27 Last patient last visit
Period: Overall Study
Arm/Group | One-day Sampling With One-year Interval | Two-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With Two-year Interval | Hp Stool Antigen (HpSA)+FIT | FIT Only
Started | 9076 | 8987 | 9032 | 8945 | 31497 | 31777
Completed | 9076 | 8987 | 9032 | 8945 | 31497 | 31777
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Average risk population
Groups:
- Total: Total of all reporting groups
Arm/Group | One-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With One-year Interval | Two-day Sampling With Two-year Interval | Hp Stool Antigen (HpSA)+FIT | FIT Only | Total
Number analyzed (Participants) | 9076 | 8987 | 9032 | 8945 | 31497 | 31777 | 99314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7248 | 7492 | 7220 | 7474 | 25393 | 25556 | 80383
  >=65 years | 1828 | 1495 | 1812 | 1471 | 6104 | 6221 | 18931
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5206 | 4941 | 5124 | 4990 | 18473 | 18523 | 57257
  Male | 3870 | 4046 | 3908 | 3955 | 13024 | 13254 | 42057
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9076 | 8987 | 9032 | 8945 | 31497 | 31777 | 99314
Gastric cancer and colorectal cancer incidence/mortality [Count of Participants; unit: Participants] | 9076 | 8987 | 9032 | 8945 | 31497 | 31777 | 99314

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Stomach Cancer
Description: Number of incident stomach cancer
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: Average risk population
Measure: Count of Participants; unit: Participants
Arm/Group | Hp Stool Antigen (HpSA)+FIT | FIT Only
Number analyzed (Participants) | 31497 | 31777
Participants | 49 | 59

2. Primary Outcome: Mortality of Stomach Cancer
Description: Number of stomach cancer death
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: Average risk population
Measure: Count of Participants; unit: Participants
Arm/Group | Hp Stool Antigen (HpSA)+FIT | FIT Only
Number analyzed (Participants) | 31497 | 31777
Participants | 17 | 23

3. Secondary Outcome: Mortality of Colorectal Cancer
Description: Number of colorectal cancer death
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: Average risk population
Measure: Count of Participants; unit: Participants
Arm/Group | One-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With One-year Interval | Two-day Sampling With Two-year Interval
Number analyzed (Participants) | 9076 | 8987 | 9032 | 8945
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Incidence of Colorectal Cancer
Description: Number of incident colorectal cancer
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: Average risk population
Measure: Count of Participants; unit: Participants
Arm/Group | One-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With One-year Interval | Two-day Sampling With Two-year Interval
Number analyzed (Participants) | 9076 | 8987 | 9032 | 8945
Participants | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: Helicobacter Pylori Eradication Rate
Description: Subjects who received anti-H. pylori treatment.
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: subjects with HpSA positive test
Measure: Count of Participants; unit: Participants
Arm/Group | Hp Stool Antigen (HpSA)+FIT
Number analyzed (Participants) | 12142
Participants | 8809

6. Other Pre Specified Outcome: Confirmatory Examination Referral Rate
Description: Subjects who received confirmatory examinations (colonoscopy or flexible sigmoidoscopy plus double contrast barium enema for lower gastrointestinal tract disease; esophagogastroduodenoscopy for upper gastrointestinal tract disease) /subjects with positive stool test (FIT or HpSA)
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: subjects with positive stool test
Measure: Count of Participants; unit: Participants
Groups:
- Hp Stool Antigen (HpSA) + FIT: HpSA for detection of upper gastrointestinal tract diseases and upper endoscopy for H. pylori carriers; HPSA combined with FIT
  HpSA (Firstep Helicobacter pylori Antigen Rapid Test): HpSA for detection of upper gastrointestinal diseases; screen and treat for H. pylori infection. Upper endoscopy for H. pylori carriers. HPSA+FIT compared with FIT alone.
Arm/Group | One-day Sampling With One-year Interval | Two-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With Two-year Interval | Hp Stool Antigen (HpSA) + FIT | FIT Only
Number analyzed (Participants) | 486 | 712 | 506 | 719 | 2230 | 2214
Participants | 328 | 473 | 355 | 493 | 1724 | 1739

7. Other Pre Specified Outcome: Detection of Advanced Adenoma and Cancer
Description: Number of Advanced Adenoma and Colorectal Cancer
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | One-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With One-year Interval | Two-day Sampling With Two-year Interval
Number analyzed (Participants) | 9076 | 8987 | 9032 | 8945
Participants | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Participation Rate of HpSA + FIT or FIT Only
Description: Number of participants from invitation population
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: Average risk population
Measure: Count of Participants; unit: Participants
Arm/Group | Hp Stool Antigen (HpSA)+FIT | FIT Only
Number analyzed (Participants) | 63508 | 88995
Participants | 31497 | 31777

9. Other Pre Specified Outcome: Detection of Non-advanced Adenoma
Description: Number of non-advanced adenoma from study population
  The recruitment period of participants was from January 1, 2014 to September 27, 2018. Final follow-up occurred December 31, 2020.
  For outcome measurement, the average follow-up time of the study participants was 5.5 years.
Time Frame: 5.5 years
Population: Average risk population
Measure: Count of Participants; unit: Participants
Arm/Group | One-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With One-year Interval | Two-day Sampling With Two-year Interval
Number analyzed (Participants) | 9076 | 8987 | 9032 | 8945
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5.5 years
Arm/Group | One-day Sampling With One-year Interval | Two-day Sampling With One-year Interval | One-day Sampling With Two-year Interval | Two-day Sampling With Two-year Interval | Hp Stool Antigen (HpSA)+FIT | FIT Only
All-Cause Mortality (participants affected / at risk) | 0/9076 | 0/8987 | 0/9032 | 0/8945 | 34/31497 | 37/31777
Serious Adverse Events (participants affected / at risk) | 0/9076 | 0/8987 | 0/9032 | 0/8945 | 0/31497 | 0/31777
Other Adverse Events (participants affected / at risk) | 0/9076 | 0/8987 | 0/9032 | 0/8945 | 0/31497 | 0/31777

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2012-05-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT01741363/Prot_000.pdf
  • Statistical Analysis Plan (2012-05-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT01741363/SAP_001.pdf
  • Informed Consent Form (2013-06-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT01741363/ICF_002.pdf